CLINICAL TRIAL: NCT04182737
Title: Efficacy and Safety of Adjunctive IgM-enriched Immunoglobulin Therapy With a Personalized Dose Based on Serum IgM-titers vs. Standard Dose in Patients With Septic Shock. A Multicenter, Interventional, Randomized, Single-blinded, Two Arms Trial.
Brief Title: Efficacy and Safety of Therapy With IgM-enriched Immunoglobulin With a Personalized Dose vs Standard Dose in Patients With Septic Shock.
Acronym: IgM-FAT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massimo Girardis (Other)
Responsible Party: Sponsor-Investigator, Massimo Girardis, Professor, University of Modena and Reggio Emilia
Organization: University of Modena and Reggio Emilia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IgM-FAT-3.0-22-12-2018; 2018-001613-33 (EudraCT Number)
Record Dates: First submitted 2019-11-26; First posted 2019-12-02 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Shock, Septic; Sepsis; Hypoglobulinemia
Keywords: immunoglobulins; septic shock; adjunctive treatment; critically ill patients
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — pentaglobulin

STUDY DESIGN:
Intervention Model Description: The study is designed as a multicentre, national, interventional, randomized, single-blinded, prospective, investigator sponsored, two arms study. Patients, who satisfy all inclusion criteria and no exclusion criteria, will be randomly assigned to IgM titer-based treatment or flat treatment group in a ratio 1:1. A block randomisation will be used with variable block sizes (block size 4-6-8), stratified by centre. Central randomisation will be performed using a secure, web-based, randomisation system. The allocation sequence will be generated by the study statistician using computer generated random numbers.
Who Masked: Participant
Masking Description: The study is conceived as single blinded: only the patients will be not aware of the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IgM titer-based treatment (Experimental): The treatment with IgM preparation will be initiated as soon as possible after randomization (maximum allowed starting time 12h after randomization). The calculation of the dose is based on IgM single compartment distribution. The first dose of IgM preparation will be calculated on IgM serum concentration obtained within 24 hours after shock appearance to achieve serum titers above 100mg/dl. In the next days, the daily IgM preparation dose will be assessed individually on the basis of IgM serum titers assessment performed in the morning with the purpose of maintaining IgM serum titers above 100 mg/dl, up to discontinuation of vasoactive drugs or day 7 after enrolment. Daily, the calculated dose will be administered in 24 hours in continuous infusion with a maximum infusion rate of 0,4 ml/kg per hour (20mg/kg per hour). IgM preparation will be administered up to the withdrawal of vasoactive drugs with a maximum allowed of 7 days of therapy and a maximum dose of 350mg/Kg/day.
  Interventions: Drug: IgM-enriched polyclonal immunoglobulins titer-based treatment
- IgM Flat treatment (Active Comparator): The IgM treatment will be initiated as soon as possible after randomization (maximum allowed starting time 12h after randomization). The dose of IgM preparation will be 250mg/kg for 3 days, the dose will be administered in 24 hours in continuous infusion with a maximum infusion rate of 0,4 ml/kg (20mg/kg per hour) until reaching 250mg/kg.
  Interventions: Drug: IgM-enriched polyclonal immunoglobulins Flat treatment

INTERVENTIONS:
Drug: IgM-enriched polyclonal immunoglobulins titer-based treatment — Immunoglobulins will be administered in a personalized dose based on serum IgM-titers
  Other Names: Pentaglobin®; IgM-enriched polyclonal immunoglobulins
  Arms: IgM titer-based treatment
Drug: IgM-enriched polyclonal immunoglobulins Flat treatment — Polyclonal endovenous immunoglobulins enriched in IgM administered in standard fixed dosages
  Other Names: Pentaglobin®; IgM-enriched polyclonal immunoglobulins
  Arms: IgM Flat treatment

SUMMARY:
In patients with septic shock, low levels of circulating immunoglobulins are common and they are kinetic, particularly of immunoglobulin M (IgM), seems to be related with clinical outcome. These observations, combined with the pivotal role of immunoglobulins on host immune response to infections, led to consider therapy with polyclonal intravenous immunoglobulins a promising option in patients with septic shock.

IgM-enriched preparations have been used since now most of all at a standard dose recommended by the producer although a more tailored approach may improve patients' outcomes.

This study hypothesizes that in patients with septic shock and low IgM immunoglobulins titers at shock onset, adjunctive treatment with a personalized dose of IgM-enriched immunoglobulins based on IgM serum titers of the patient may reduce mortality compared to a standard dose of IgM-enriched immunoglobulins. The study is designed as a multicentre, national, interventional, randomized, single-blinded, prospective, investigator-sponsored, two arms study. Patients will be randomly assigned to IgM titer-based treatment or flat treatment group in a 1:1 ratio. One group of patients will receive IgM-enriched immunoglobulins adjunctive treatment in a standard dose of 250mg/kg for 3 days. The other group will receive IgM-enriched immunoglobulins adjunctive treatment in a variable dose calculated taking note of the extent of IgM deficit, in order to achieve an IgM threshold value of 100 mg/dL or above. IgM preparation will be administered in this group up to the withdrawal of vasoactive drugs with a maximum allowed of 7 days. The confirmation of the efficacy of a tailored strategy for IgM-enriched immunoglobulin administration in reducing the mortality rate among patients with septic shock and low IgM titers will lead to a revision of the current clinical practice in the use of this adjunctive treatment.

DETAILED DESCRIPTION:
Rationale:

Several clinical studies have reported that serum immunoglobulins concentrations are generally low in patients with sepsis and that the level and kinetics of serum immunoglobulins, particularly immunoglobulin M (IgM), seem to be somehow related to patient outcome. Intravenous administration of immunoglobulin preparations seems to be a promising treatment option due to their pleiotropic effects on bacteria and the host response to infections.

In previous clinical experiences, IgM preparation has been mainly administered at the dosage recommended by Summary of Product Characteristics (250 mg/Kg/day for three consecutive days) regardless of the patient severity and without any adjustment based on immunoglobulins plasma concentration or other biomarkers. The recent understanding of the high heterogeneity in pathobiology led to recommend a more tailored approach in patients with sepsis by modulating therapies on the basis of specific clinical and biological markers. Therefore, nowadays the strategy of a fixed-dose should be revised.

Our study hypothesis is that a personalized administration of IgM-enriched immunoglobulin, calculated based on serum IgM-titers of the patient, will decrease mortality compared to standard IgM-enriched immunoglobulin treatment (fixed or flat dose).

Study objective:

The primary objective is to verify the hypothesis that adjunctive therapy with IgM-enriched immunoglobulin with a personalized dose based on serum IgM-titers is more effective in reducing any-cause mortality in patients with septic shock compared to a flat dose therapy. Mortality will be measured at 28 days.

The confirmation of the efficacy of an IgM-titre based dose of IgM preparation reducing the mortality rate among patients with septic shock will lead to a revision of the current clinical practice in the use of this adjunctive therapy.

Study setting:

The study will involve 12 Italian Intensive Care Units (ICUs). The recruitment of 356 participants will be completed in around 24 months.

Interventions:

Patients who satisfy all inclusion criteria and no exclusion criteria will be randomly assigned to an IgM titer-based treatment group (Group 1) or an IgM Flat treatment group (group 2) in a ratio1:1.

The treatment given to patients of both groups during this independent study will be the IgM-enriched immunoglobulin preparation (IgM preparation) (Pentaglobin®, Biotest, Germany) commercially available. The IgM preparation contains high titers of antibodies against lipopolysaccharides and outer membrane proteins of many Gram-negative bacteria. Composition active ingredients: 1 ml solution contains Human plasma protein 50 mg of which immunoglobulin at least 95 %, IgM 6 mg, immunoglobulin A (IgA) 6 mg, immunoglobulin G (IgG) 38 mg. Other constituents: Glucose monohydrate (27.5 mg/ml), sodium chloride (78 μmol/ml), water for injections (ad 1 ml).

Group 1 (IgM titer-based treatment): The treatment with IgM preparation will be initiated as soon as possible after randomization (maximum allowed starting time 12h after randomization). The calculation of the dose is based on IgM single compartment distribution. The first dose of IgM preparation will be calculated on IgM serum concentration obtained within 24 hours after shock appearance to achieve serum titers above 100mg/dl. In the next days, the daily IgM preparation dose will be assessed individually on the basis of IgM serum titers morning assessment, with the purpose of maintaining IgM serum titers above 100mg/dl, up to discontinuation of vasoactive drugs or day 7 after enrolment. If the serum titer is above 100 mg/dl, the daily dose of IgM-preparation will be zero, up to the daily serum titer decreases below 100 mg/dl. In this case, the patient will remain in the study despite he will not receive the daily dose of IgM preparation. If for whatever reason, IgM serum titers result is not available, the daily dose will be calculated using the last IgM result obtained within 48 hours. The threshold of 100 mg/dl of IgM serum titers is based on internal preliminary unpublished data from the University Hospital of Modena showing protective effects compared to lower levels of IgM. Daily, the calculated dose will be administered in 24 hours in continuous infusion with a maximum infusion rate of 0,4 ml/kg per hour (20mg/kg per hour) until reaching the calculated daily dose.

IgM preparation will be administered up to the withdrawal of vasoactive drugs with a maximum allowed of 7 days of therapy and a maximum dose of 350mg/Kg/day, as reported from previous experiences.

Group 2 (IgM Flat treatment): The IgM treatment will be initiated as soon as possible after randomization (maximum allowed starting time 12h after randomization). The dose of IgM preparation will be 250mg/kg for 3 days, the dose will be administered in 24 hours in continuous infusion with a maximum infusion rate of 0,4 ml/kg (20mg/kg per hour) until reaching 250mg/kg.

In both groups, before enrolment in the study, it will be allowed the administration of intravenous immunoglobulins (either Immunoglobulin G or IgM-enriched preparation) at standard dosages for a maximum of 6 hours.

Concomitant medications:

Depending on their clinical status, patients will be treated according to the principles of the Good Clinical Practice, Survival Sepsis guidelines 2016 and clinical judgement of the attending physician. No other pharmacological therapy or treatment will be influenced by the study protocol. There are no restrictions to concomitant treatments provided to patients in this study. All relevant concomitant medications and treatments took or administered in the 24 hours before the screening and during the study period will be recorded.

Criteria for discontinuing or modifying allocated interventions:

The duration of study therapy will be until the withdrawal of vasoactive drugs with a maximum allowed of 7 days of therapy in the IgM titer based group and 3 days in the Flat treatment group.

Patients may be prematurely discontinued from study protocol at the discretion of the Investigator, should any untoward effect occur (including an adverse event (AE) or clinically significant laboratory abnormality that, in the opinion of the Investigator, warrants the subject's permanent discontinuation of study protocol-directed care).

Data collection and management:

Every patient who meets the inclusion criteria will be included and randomised in the two groups. The study data will be collected along the entire study period in a dedicated electronic Case Report Form (eCRF). The eCRF will be provided by the steering committee with proper options to minimize data entry errors: the data will incorporate un-amendable fixed intervals of values (for continuous variables) and pre-defined coding system (for binary or categorical variables). Data entry will be performed and double-checked from a dedicated researcher in each centre; in order to limit collection errors, records will be randomly re-checked from the PI. The data collection will be also checked by a Clinical Monitor, assigned by the contract research organization (CRO), by phone calls and visits at the study sites as agreed with the investigators. The study Monitor will be responsible for performing the monitoring in accordance with good clinical practice (GCP) guidelines. The investigators and the CRO will agree on monitoring visits to assess the progress of the study, verify adherence to the protocol, check the eligibility of patients, the accuracy and completeness of the eCRF, check the correlation between the data reported into eCRF and those recorded in the hospital documents (medical records, patient registries, etc.), check for the correct reporting of adverse events, verify that evaluations planned and documentation of the study are properly stored and handled.

All the data about the included patients will be extrapolated from the clinical documentation and recorded in an eCRF from the adequately trained researcher. Demographic information (gender, age), co-morbidities, reason of ICU admission, type of ICU admission (medical, elective surgery, emergency surgery) will be registered at the inclusion, severity of critical illness quantified by the Simplified Acute Physiology Score II (SAPS II) will be calculated by the data from the first 24 h of ICU stay. During the study duration clinical and laboratory parameters will be evaluated and recorded following the scheduled times: IgM titers, simplified organ failure assessment (SOFA) score and its components, Multiple Organ Failure score (MOF score) and its components, vital signs such as mean arterial pressure, heart rate, respiratory rate, systemic temperature, diuresis, fluid balance, data from routine laboratory test such as haemoglobin, platelets count, white blood cells count, troponin, coagulative parameters, parameters for liver and renal function, oxygen inspired fraction, blood gas analysis results, ventilation mode, need of renal replacement therapy, blood cells count, C-reactive protein, procalcitonin, occurrence of ICU-acquired blood, respiratory and urinary-tract infection and the implicated microorganisms, reactivation of viral infections and MRC scale.

Other recorded parameters will include the duration of ventilatory support in days, duration and type of antibiotic and antifungal therapy in days, need and the dose of vasoactive drugs.

The application of evidence-based treatments recommended by the guidelines (i.e. blood collection for microbiological culture, antibiotic and fluid therapies, and the eventual use of specific adjunctive therapies as for instance steroids and blood purification) will be recorded.

As a blood-bank for possible further biochemical investigations (e.g. cytokines titers, different biomarkers), for each patient who will be included in the study a blood sample of about 6 ml will be collected at baseline, day 7 and 28 or ICU discharge and stored, after centrifugation, at -70°C in the local laboratory of each site.

Methods for statistical analysis The intention to treat population will be considered for the primary analysis. A descriptive statistical analysis will be performed to describe every relevant variable. Kolmogorov-Smirnov normality test will be performed in order to verify the distribution of the variables. Baseline variables will be compared between the two groups using the Mann-Whitney U test or t-test as appropriate. Categorical variables will be compared using Fisher's Exact test. The primary outcome will be assessed by comparison of proportions of patients alive in both groups at day 28 by using Fisher's exact test. To compare the treatment effect on the secondary outcomes will be assessed as follow: all-cause of mortality at ICU discharge, at hospital discharge and at day 90 by Fisher's exact test; occurrence of new organ dysfunctions and grade or dysfunctions in all the study period by Fisher's exact test and distribution-free test such as median test respectively; intensive care unit free hours (IFHs) at 28-day, hospital free days (HFDs) at day 90, ventilator-free days (VFDs) at 28-day, vasopressors free days (VasoFDs) at 28-day, antibiotic-free days (AFDs) at 28-day by distribution-free test such as median; ICU acquired weakness assessed with Medical Research Council (MRC) Scale for Muscle Strength by analysis of variance including terms for treatment, time and centre.

Every test will be performed considering a two-sided p-value < 0,05 for statistical significance. In general, categorical data will be presented using counts and percentages, whilst continuous variables will be presented using the number of patients, mean, standard deviation, median, minimum, and maximum. 95% confidence interval will be calculated for the primary variable and the relevant secondary variables.

Subgroup analysis: The primary and secondary outcomes will be evaluated in pre-defined subgroups: distribution of SAPS II and SOFA score (total and for single organ) at admission, surgical admissions compared to non-surgical admissions, type of pathogen cause of septic shock, site and type of infection, distribution of IgM and IgG plasma concentration at baseline and at day 3, biomarkers reactive protein C (CRP) and procalcitonin (PCT) distribution at baseline and at day 3, patients with end-stage liver disease compared to patients without and patients with malignancies compared to patients without.

Data monitoring An independent Data Safety Monitoring Board (DSMB), consisting of 2 experts in clinical research in intensive care and 1bio-statistic will be established before patient enrolment. The DSMB Charter will be prepared by the steering committee and signed by the members of the DSMB before the trial commences. The DSMB will have access to all results and make the appropriate considerations about the appropriateness of the sample size, the efficiency and quality of data collection system, eventual occurrence of a suspected protocol-related adverse event. The DSMB has the right to stop the trial for safety reasons.

Analyses ad interim Considering a statistical approach based on two phases, an interim analysis is planned after the randomization of 178 patients (50% of sample size) for the double objective of monitoring safety and verifying the accuracy of the assumptions made for sample size estimation regarding the primary end-point event rate in relation to the anticipated survival benefit. With the interim analysis, we will be able to evaluate whether there is a substantial superiority of one treatment. The obtained results will be evaluated by the DSMB and by the steering committee and, in case of significant differences in survival among the two groups, all patients will be switched to the most promising treatment.

Harms Previous studies did not identify specific risks correlated to intravenous immunoglobulins preparations enriched with IgM. However, all the included patients will be intensively monitored following the standard procedures of intensive care medicine and any suspected protocol-related adverse event will be reported to the steering committee, the data safety and monitoring board, other participating centres and the competent authorities. In Beyond suspected protocol-related adverse event, the data safety and monitoring board will have access to all results of the trial and make the appropriate considerations about the appropriateness of the sample size, the efficiency and quality of data collection system and has the right to stop the trial for safety reasons or futility.

Ethics and dissemination The study will be conducted in line with the protocol, the Declaration of Helsinki (1964) and subsequent amendments and updates(Fortaleza, Brazil, October 2013). Moreover, it is the responsibility of the investigator to ensure that the study will be done in line with the requirements of Good Clinical Practice(GCP) and the applicable regulatory requirements.

Research ethics approval The entire study protocol, including informative material for the patients and modules for the informed consent, ill be evaluated by the Local Ethics Committee (EC) from the coordinating centre and all the collaborating centres. The study will not start before obtaining a favourable opinion from the EC, the Competent Authority Authorization and any other authorization required by local regulation. Every intention to modify any element of the original protocol after the first approval will be promptly notified to the Ethics Committee and will be applied only after its written authorization.

Investigator/sponsor will be responsible to submit to the Ethics Committee any amendments to the protocol.

Consent and confidentiality Before inclusion in the study, conscious patients must be informed of the purpose and clinical procedures required by the protocol. The investigators will explain the purpose, risks and benefits associated with study participation. Besides, patients will be informed of his right to withdraw from the study at any time without explanation and without losing the right to future medical care.

If the patient will be unable to comprehend or to give his consent (because of compromised neurological status), the following consent options are acceptable: (i) A priori consent by a legal representative (ii) delayed consent from a legal representative; (iii) Delayed consent from the patient; (iv) waiver of consent; (v) consent provided by an ethics committee or other legal authority. Which options are available at individual participating sites will be determined by the relevant ethics committee and subject to applicable laws. All participants who recover sufficiently will be allowed to provide informed consent for ongoing study participation and the use of data collected for the study. Every patient is free to leave the study protocol at any stage of the study and can request to retire his consent and, consequently, to ask the elimination of all his data from the database.

In order to comply with legal requirements regarding privacy and the processing of sensitive personal data, Legislative Decree 30/06/2003 n. 196 on the protection of personal data and Regulation (EU) 2016/679 of the European Parliament and of the Council of 27 April 2016 on the protection of natural persons with regard to the processing of personal data and on the free movement of such data, and repealing Directive 95/46/EC (General Data Protection Regulation), each patient will be given an information sheet on the study they participate in and will be asked for sign the consent to the processing of personal data.

Data about personal and private information, included sensible data, will be treated following current legislation on data protection; patients will be identified with a coding system and data registered in an anonymous form. Collected data will be processed by the Investigator for the exclusive purposes of fulfilling to the present study requirements, and in an anonymous form, aggregate in the study database with data obtained from the other patients participating, solely on the basis of finalizing the study and achievement objectives.

Obtained data will not be disclosed except in strictly anonymous and aggregated form. Direct access to the original medical records may be requested only by commissioning DSMB of the study and will be accessible by a representative of the CRO, its delegate to perform monitoring on the conduct of the trial, the EC or by the Regulatory Authorities, such as personnel of the Italian Ministry of Health and the Italian Medicines Agency (AIFA) to verify that the information entered in the documents of the study is correct and methods that guarantee the privacy and confidentiality of the data are respected.

Dissemination policy The Circ. Min. Health N° 6 of 09/02/2002 obliges each researcher who gets any results of interest to public health, to publish the results within 12 months from the end of the study. All the patients will freely agree or disagree to participate in the study in the belief that the results will be useful to improve knowledge about their pathologies, for health benefit from themselves or other patients. To respect their will and in the maximum interest of honest clinical research, the investigators agree on the need to ensure the wide publication and diffusion of their results in a consistent and responsible way under their responsibility. The study coordinator is the official data owner. The steering committee has the right to present methods and results of the study at public symposia and conferences. The principal publications from the trial will be in the name of Investigators with full credit assigned to all collaborating investigators and institutions.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years;
2. Septic shock occurrence < 24 hours; septic shock is identified according to Sepsis-3 definition by a vasopressor requirement to maintain a mean arterial pressure of 65 mm Hg or greater and serum lactate level greater than 2 mmol/L (>18 mg/dL) in the absence of hypovolemia in patients with sepsis2. Sepsis is defined as a life threatening organ dysfunction identified as an acute change in total SOFA score ≥2 points consequent to the infection;
3. IgM-titers< 60mg/dl (or < 20% of the lower threshold value of local laboratory) within24hours from shock occurrence.

Exclusion Criteria:

1. Shock of uncertain diagnosis;
2. Hypersensitivity to IgM Preparation in use or its excipients;
3. Patients receiving intravenous immunoglobulins (e.g. IgG or IgM enriched preparations) for > 6 hours before enrolment;
4. Selective absolute IgA deficiency with antibodies to IgA;
5. Pregnancy or breastfeeding or positive pregnancy test. In childbearing age women, before inclusion, a pregnancy test will be performed if not available;
6. Clinical decision to withhold life-sustaining treatment or "too sick to benefit";
7. Neutrophil count <1.000/mm3;
8. Presence of other severe diseases impairing life expectancy (e.g. patients are not expected to survive 28 days given their pre-existing medical condition);
9. Patients with a known, chronic kidney dysfunction needing dialysis (creatinine ≥ 3.4 mg/dl or creatinine clearance ≤ 30 ml/min/1.73m2);
10. Body Mass Index (BMI) >40;
11. Participation in other clinical trials on adjunctive therapies for sepsis (during past 3 months);
12. Lack of withdrawal of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality at day 28 | Day 28 from randomization
  All-cause mortality at day 28, defined as the comparison of proportions of patients death for any cause at day 28 from randomization.

SECONDARY OUTCOMES:
All-cause mortality at ICU discharge | ICU discharge, censored at day 28
  All-cause mortality at ICU discharge, defined as the comparison of proportions of patients death for any cause at ICU discharge.
All-cause mortality at hospital discharge | Hospital discharge, censored at day 90
  All-cause mortality at Hospital discharge, defined as the comparison of proportions of patients death for any cause at hospital discharge
All-cause mortality at day 90 | Day 90 from randomization
  All-cause mortality at day 90, defined as the comparison of proportions of patients death for any cause at day 90
New organ dysfunction during ICU stay | From randomization to ICU discharge, censored at day 28
  Occurrence of new organ dysfunction during ICU stay. Organ dysfunction is defined as a Sequential Organ Failure Assessment (SOFA) score ≥3 for the corresponding organ occurring after randomization. SOFA score ranges from 0 (no organ dysfunction) to 24 (multiple organ failure)
New organ dysfunction during ICU stay | From randomization to ICU discharge, censored at day 28
  Occurrence of new organ dysfunction during ICU stay. Organ dysfunction is defined as a Multiple organ Failure (MOF) score ≥1 for the corresponding organ occurring after randomization. MOF ranges from 0 (no organ dysfunction) to 14 (multiple organ dysfunction)
Grade of organ dysfunction during ICU stay | From randomization to ICU discharge, censored at day 28
  Grade of organ dysfunction during ICU stay, grade of dysfunction is measured with Sequential Organ Failure Assessment (SOFA) score and with Multiple organ Failure (MOF) score daily from randomization to day 28 or ICU discharge.
ICU free hours at day 28 | From randomization to day 28
  Total number of hours between ICU discharge and day 28. If death occurs during the ICU stay before day 28 the ICU free hours calculation will be 0. The ICU readmission before day 28 after randomization will be considered.
Hospital free days at day 90 | From randomization to day 90
  Total number of days between Hospital discharge and day 90. If death occurs during the hospital stay before day 90 the hospital free days calculation will be 0. Hospital readmissions before day 90 after randomization will be considered.
Ventilation free days at day 28 | From randomization to day 28
  Total number of days that patient is alive and free of ventilation between randomisation and day 28. Periods of assisted breathing lasting less than 24 hours for surgical procedures will not count against the ventilation free days calculation.
Vasopressors free-days at day 28 | From randomization to day 28
  Total number of days that patient is alive and free of vasopressors between randomisation and day 28.
Antibiotic free days at day 28 | From randomization to day 28
  Total number of days that the patient is alive and free of antibiotic drugs administration between randomisation and day 28.
ICU acquired weakness | Day 7, 28 and 90 censored at hospital discharge
  ICU acquired weakness is defined by Medical Research Council (MRC) scale, when weakness had developed after ICU admission, is symmetric and the average MRC score is <4
Occurrence of protocol related adverse events | From randomization to day 28
  Adverse events occurred from randomization to day 28. Events that are part of the natural history of the primary disease process or expected complications of critical illness will not be reported as adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- ICU- University Hospital Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Biagioni E, Tosi M, Berlot G, Castiglione G, Corona A, De Cristofaro MG, Donati A, Feltracco P, Forfori F, Fragranza F, Murino P, Piazza O, Tullo L, Grasselli G, D'Amico R, Girardis M. Adjunctive IgM-enriched immunoglobulin therapy with a personalised dose based on serum IgM-titres versus standard dose in the treatment of septic shock: a randomised controlled trial (IgM-fat trial). BMJ Open. 2021 Feb 11;11(2):e036616. doi: 10.1136/bmjopen-2019-036616. PMID 33574139